CLINICAL TRIAL: NCT01073826
Title: A Lifestyle Intervention Study Investigating the Role of Interleukin-6 in the Beneficial Effect of Exercise on Beta-cell Function in Obese People and Patients With Type 2 Diabetes
Brief Title: Role of Interleukin-6 in Exercise
Acronym: Exil-6
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: European Foundation for the Study of Diabetes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Donath-1
Record Dates: First submitted 2009-10-19; First posted 2010-02-23 (Estimated); Last update posted 2016-11-01 (Estimated); Status verified 2016-10

CONDITIONS: Diabetes Mellitus, Type 2; Obesity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity | interventions — tocilizumab; Sitagliptin Phosphate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Tocilizumab (Active Comparator): Infusion of Tocilizumab and sport intervention
  Interventions: Behavioral: Sport; Drug: Tocilizumab
- Sitagliptin (Active Comparator): Intake of Sitagliptin and sport intervention
  Interventions: Behavioral: Sport; Drug: Sitagliptin
- Placebo (Placebo Comparator): Intake of placebo and sport intervention
  Interventions: Behavioral: Sport

INTERVENTIONS:
Behavioral: Sport
Drug: Tocilizumab
  Arms: Tocilizumab
Drug: Sitagliptin
  Arms: Sitagliptin

SUMMARY:
The purpose of the study is to understand the role of interleukin-6 during physical activity in patients with type 2 diabetes.

ELIGIBILITY:
Inclusion criteria:

* Obesity group: BMI 30-40 kg/m2, fasting plasma glucose <6.4 mmol/l.
* Diabetes group: Type 2 diabetes according to American Diabetes Association criteria

Exclusion criteria:

* Anti-diabetic drug other than metformin
* Diabetes duration of more than 5 years
* Inflammatory diseases
* Current infection
* Liver disease (transaminases >2x upper normal range)
* kidney disease (creatinine >1.5 mg/dl for men and 1.4 mg/dl for women)
* pregnancy or breast-feeding, women of child bearing potential not using an acceptable form of contraception
* immunosuppressive disease
* corticosteroid use
* regular non-steroidal antinflammatory drug usage
* history of carcinoma
* history of tuberculosis
* anemia, bleeding disorders
* obstructive pulmonary disease.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2010-02; Primary Completion 2015-11 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Glucagon like peptide- 1 (GLP-1) | Change in GLP-1 secretion compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: 01 Studienregister MasterAdmins, Study Director — UniversitaetsSpital Zuerich
Locations (1):
- University Hospital Zurich, Zurich, Switzerland

REFERENCES:
- [Derived] Ellingsgaard H, Seelig E, Timper K, Coslovsky M, Soederlund L, Lyngbaek MP, Wewer Albrechtsen NJ, Schmidt-Trucksass A, Hanssen H, Frey WO, Karstoft K, Pedersen BK, Boni-Schnetzler M, Donath MY. GLP-1 secretion is regulated by IL-6 signalling: a randomised, placebo-controlled study. Diabetologia. 2020 Feb;63(2):362-373. doi: 10.1007/s00125-019-05045-y. Epub 2019 Dec 3. PMID 31796986